CLINICAL TRIAL: NCT03379974
Title: Exercise Versus DDAVP in Patients With Mild Hemophilia A - is One Non-inferior to the Other and do They Work Additively in Improving Hemostasis?
Brief Title: Exercise Versus DDAVP in Patients With Mild Hemophilia A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-00290
Record Dates: First submitted 2017-12-05; First posted 2017-12-20 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Masking Description: The randomization of the participant to a study arm will be done prior to the study visit by the pharmacy at the hospital. The Investigator and study team will know the arm each participant is in before the patient's visit. This information will also be provided to the participant before the visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ARM A: DDAVP followed by exercise (Experimental): 1. Intervention #1: DDAVP Inhalant Product intervention The participant will take either 1 or 2 nasal sprays of IN DDAVP. For patients weighing <50 kg: 150 ug (i.e. 1 spray into one nostril) and patients weighing ≥50 kg: 300 ug (i.e. 2 sprays - one into each nostril).
  2. Intervention #2: Exercise intervention
  Interventions: Drug: DDAVP Inhalant Product; Behavioral: Exercise Intervention
- ARM B: DDAVP alone (Active Comparator): 1. Intervention #1: DDAVP Inhalant Product intervention The participant will take either 1 or 2 nasal sprays of IN DDAVP. For patients weighing <50 kg: 150 ug (i.e. 1 spray into one nostril) and patients weighing ≥50 kg: 300 ug (i.e. 2 sprays - one into each nostril).
  2. Intervention #2: no further intervention (rest)
  Interventions: Drug: DDAVP Inhalant Product
- ARM C: Exercise intervention (Experimental): 1. Intervention #1: Exercise intervention
  2. Intervention #2: no further intervention (rest)
  Interventions: Behavioral: Exercise Intervention
- ARM D: Exercise followed by DDAVP (Experimental): 1. Intervention #1: Exercise intervention
  2. Intervention #2: DDAVP Inhalant Product intervention The participant will take either 1 or 2 nasal sprays of IN DDAVP. For patients weighing <50 kg: 150 ug (i.e. 1 spray into one nostril) and patients weighing ≥50 kg: 300 ug (i.e. 2 sprays - one into each nostril).
  Interventions: Drug: DDAVP Inhalant Product; Behavioral: Exercise Intervention

INTERVENTIONS:
Drug: DDAVP Inhalant Product — For the DDAVP intervention the participant will take either 1 or 2 nasal sprays of IN DDAVP. After receiving IN DDAVP, the participant will rest for 30 minutes.
  Other Names: IN DDAVP
  Arms: ARM A: DDAVP followed by exercise; ARM B: DDAVP alone; ARM D: Exercise followed by DDAVP
Behavioral: Exercise Intervention — For the exercise intervention the participant will exercise on a stationary cycle-ergometer using the previously-validated, progressively-incremental Godfrey protocol. Per the Godfrey protocol, the participant starts cycling on the calibrated cycle-ergometer with an initial exercise load that is dependent on their height. The workload is increased every minute in standard increments also based on the participant's height. All participants will exercise till they complete 3-minutes of cycling at 85% of their maximum predicted heart rate or till exhaustion (whichever comes first). Upon completion of planned exercise, work load will be decreased to zero watts and participants will be instructed to continue cycling at this cool-down rate for additional 3-minutes, before getting of the ergometer.
  Arms: ARM A: DDAVP followed by exercise; ARM C: Exercise intervention; ARM D: Exercise followed by DDAVP

SUMMARY:
Individuals with mild hemophilia A (MHA) bleed infrequently but can in the setting of trauma which often is when participating in sports/exercise. Although both exercise and DDAVP (desmopressin) can raise Factor 8/Von Willebrand Factor (FVIII/VWF levels), it is not clear whether the pathophysiological mechanism is the same. Consequently it is not known if DDAVP and exercise would have additive effects in raising FVIII:C and VWF levels or if one would one negate the effect of the other. The aim of this 2 center (Sickkids and Nationwide Children's), prospective, cross-over design study is to compare the impact of exercise vs. DDAVP on hemostasis in patients with MHA and also to investigate the impact of sequentially administering these interventions on their hemostatic indices.

DETAILED DESCRIPTION:
Persons with mild hemophilia A (MHA) (defined as having a FVIII level of >5% to ≈50%) bleed infrequently but can in the setting of trauma which can often is in the context of participating in sports/exercise. FVIII levels temporarily rise with stress, exercise and with DDAVP (1-desamino-8-Darginine vasopressin, desmopressin). In the case of DDAVP, the Hospital for Sick Children (SickKids) Hemophilia Team and others have shown that FVIII and VWF levels rise by 2-4 fold with DDAVP. Consequently many persons with MHA in an attempt to reduce their risk of bleeding take intranasal (IN) DDAVP prior to sports activities/exercise. IN DDAVP is reasonably expensive ($300/bottle of Octistim® in Canada and $700/bottle of Stimate® in USA), requires fluid restriction, and may be associated with nausea, vomiting, seizures and tachyphylaxis.

Recently, our group completed a pilot/feasibility study to evaluate the impact of a prescribed, moderate intensity aerobic exercise regimen on hemostatic indices in 30 children with hemophilia A [HA] or B [HB] (all severities) and documented a significant improvement in multiple coagulation parameters (platelet count, FVIII:C and von Willebrand factor [VWF]) with exercise. This improvement was particularly pronounced in 13 post-adolescent males with mild-moderate HA. In this sub-cohort, the investigators noted a mean 2.3 fold increase in FVIII:C immediately after exercise, which remained significantly elevated at 1.9 fold,1 hour after completion of exercise

These changes in hemostatic variables associated with aerobic exercise may be protective against bleeding, and may negate the need to administer IN DDAVP immediately prior to sports participation.

Although both exercise and DDAVP can raise FVIII/VWF levels, it is not clear whether the pathophysiological mechanism in which they do this is the same. Consequently it is not known if DDAVP and exercise would augment each other's effects in raising FVIII:C and VWF levels or if one would one negate the effect of the other. Herein, the investigators propose a prospective, interventional study of exercise vs IN DDAVP in 40-50 post adolescent (13-21 yr) males with MHA to compare their impact on hemostasis and also to investigate the impact of sequentially administering these interventions on hemostatic indices.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients of ≥13 years of age and ≤21 years of age with MHA (FVIII:C level of ≥6% to ≤50%).

Exclusion Criteria:

1. A currently circulating or a history of inhibitor (0.5 BU on two or more occasions). Inhibitor development is rare in MHA.
2. History of FVIII infusion (both standard-acting and extended half-life products) or DDAVP use in preceding 1 week. Patients will be instructed to hold factor use or DDAVP for 1-week prior to participation in study, except for management of acute bleeds, in which case they will be instructed to inform the PI via telephone or e-mail.
3. Patients with severe arthropathy (as determined by the principal investigator) interfering with ability to exercise. Severe arthropathy is rare in MHA.
4. Patients on beta-blockers, anti-platelet agents or regular non-steroidal anti-inflammatory medications (e.g. Celebrex).
5. Patients who are active smokers (cigarettes, marijuana).
6. Patients with a history of a recent bleed (in preceding 2 weeks) in any location or a joint/muscle bleed in the lower limbs in the preceding 4 weeks.
7. Co-existence of a congenital bleeding disorder other than MHA (e.g. VWD).
8. Patients with an active infectious or inflammatory condition. This includes previously identified HIV, active hepatitis B or C as reflected in elevated AST, ALT, RNA positivity for hepatitis B or C. HIV, hepatitis B and C are very rare in the age group (13-21 years) we hope to accrue in the proposed study.
9. Patients who for medical reasons should not receive DDAVP [those with renal or CNS disease (e.g. brain tumor)] or have previously experienced adverse events with DDAVP (e.g. hypotensive event, seizure).

Ages: 13 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
•Factor 8 level after exercise [ Time Frame: Baseline, 30 min post intervention #1, 30 min post intervention #2 and 90 minute post intervention #2 | Baseline, 30 min post intervention #1, 30 min post intervention #2 and 90 minute post intervention #2
  To compare the increase in FVIII:C (measured as absolute and fold increase) associated with a standardized moderate intensity aerobic exercise regimen (3-minutes of exercise at 85% of the predicted maximum heart rate) to intranasal DDAVP in post-adolescent males with MHA

SECONDARY OUTCOMES:
•Factor 8 level after sequential administration of exercise followed by IN DDAVP (or vice versa) [ Time Frame: Baseline, 30 min post intervention #1, 30 min post intervention #2 and 90 minute post intervention | Baseline, 30 min post intervention #1, 30 min post intervention #2 and 90 minute post intervention
  To determine the absolute and fold increase in FVIII:C associated with the sequential administration of exercise followed by intranasal DDAVP (or vice versa)
•Associations between baseline physical activity scores and Factor 8 levels after exercise [ Time Frame: Baseline, 30 min post intervention #1, 30 min post intervention #2 and 90 minute post intervention | Baseline, 30 min post intervention #1, 30 min post intervention #2 and 90 minute post intervention
  To explore the impact of baseline physical activity (measured using the International Physical Activity Questionnaire [IPAQ]-short form) on exercise induced increase in FVIII:C

CONTACTS AND LOCATIONS:
Overall Officials: Riten Kumar, MD, MSc, Principal Investigator — Nationwide Children's Hospital
Locations (4):
- United States (4):
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - Akron Children's Hospital, Akron, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: Yes
To ensure the safety of patients and to confirm the validity of our hypothesis, we plan to:
  * Meet after the first 10 patients have completed the study.
  * Analyze data from first 10 patients. This includes safety data as well as results of the blood tests including the standard hemostasis testing (FVIII;C, VWF:Ag, VWF:RCo, VWF:CBA, VWF:pp), platelet function (PFA), Thromboelastography (TEG) and Thrombin generation.
  * Determine whether there are measurable outcomes justifying further enrollment and DSMB will be able to make recommendations regarding terminating the study or amending the protocol if they deem that there are safety issues.
  If any of the first 10 subjects develops any unexpected medical complication we will suspend recruitment pending re-evaluation of the study by the DSMB.